CLINICAL TRIAL: NCT00341133
Title: Genetic Analysis of Left-Right Axis Malformations
Brief Title: Genetic Analysis of Left-Right Axis Formations
Status: Completed | Type: Observational
Sponsor: National Human Genome Research Institute (NHGRI) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 999999054; OH99-HG-N054
Record Dates: First submitted 2006-06-19; First posted 2006-06-21 (Estimated); Last update posted 2017-07-02 (Actual); Status verified 2009-08-04

CONDITIONS: Congenital Heart Disease
Keywords: Laterality; Heterotaxy; Holoprosencephaly; Genetic Testing; Congential Cardiac Malformations; Disturbed Internal Organ Positioning
MeSH Terms: conditions — Heart Defects, Congenital; Situs Inversus; Holoprosencephaly

SUMMARY:
The objective of these studies is to identify genetic factors that contribute to the pathogenesis of complex congenital heart disease and other more rare conditions resulting from disturbances in organ positioning. These are a group of medical conditions that are thought to stem from a poorly understood disturbance in the establishment of the basic body plan in the embryo. While the outside of the human body is generally symmetric with mirror image left and right sides, the positions of some internal organs are distinctly asymmetric. For example, the heart could not function properly as a mechanical pump if its connections to major blood vessels retained their initial symmetry. The left ventricle of the heart normally pumps blood to the body, while the right ventricle normally pumps blood to the lungs. Reversals in these blood vessel connections can be fatal. Similarly, the gut characteristically loops in a counterclockwise direction placing the stomach on the left side in most cases. Rare laterality anomalies can occur if this looping is in the other direction, or randomized (equally likely to loop in either direction). Serious medical problems can be caused by disturbances in the establishment, or maintenance of left-right (L-R) differences as key organs are developing in the embryo.

We have established formal collaborative agreements with three major centers who have collected a large number of coded cases of congenital cardiac disease. Our research objective is to try to understand if specific genetic changes can contribute to a range of cardiac malformations. We utilize mutational analysis of candidate genes as our principal tool to study the genetics of L-R axis malformations. This protocol is also open to other conditions whose basis is also thought to result from L-R problems. In all cases, the patients continue under the care of the referring physician. We anticipate a minor role of NIH researchers and genetic counseling services if subjects either do not have, or cannot afford, similar services in their local area.

This is not a treatment protocol. Our empiric ability to generate medically significant research results is limited by the extensive genetic and other etiologic heterogeneity. Therefore, this research is not a diagnostic study. At this stage of research, we are not sufficiently confident that our research results will have direct medical implications for research subjects.

Results that are of potential medical importance will be discussed with the primary physician who is (in most cases) a trained cardiologist (and/or medical geneticist). We will emphasize that these are only preliminary research findings, that they are not CLIA-approved, and must be disclosed to the patient or included in the medical record. Repeat testing in a CLIA-approved lab under another protocol would be required before the genetic information could be shared with the patient and family.

DETAILED DESCRIPTION:
The objective of these studies is to identify genetic factors that contribute to the pathogenesis of complex congenital heart disease and other more rare conditions resulting from disturbances in organ positioning. These are a group of medical conditions that are thought to stem from a poorly understood disturbance in the establishment of the basic body plan in the embryo. While the outside of the human body is generally symmetric with mirror image left and right sides, the positions of some internal organs are distinctly asymmetric. For example, the heart could not function properly as a mechanical pump if its connections to major blood vessels retained their initial symmetry. The left ventricle of the heart normally pumps blood to the body, while the right ventricle normally pumps blood to the lungs. Reversals in these blood vessel connections can be fatal. Similarly, the gut characteristically loops in a counterclockwise direction placing the stomach on the left side in most cases. Rare laterality anomalies can occur if this looping is in the other direction, or randomized (equally likely to loop in either direction). Serious medical problems can be caused by disturbances in the establishment, or maintenance of left-right (L-R) differences as key organs are developing in the embryo.

We have established formal collaborative agreements with three major centers who have collected a large number of coded cases of congenital cardiac disease. Our research objective is to try to understand if specific genetic changes can contribute to a range of cardiac malformations. We utilize mutational analysis of candidate genes as our principal tool to study the genetics of L-R axis malformations (e.g. denaturing high performance liquid chromatography, dHPLC, or similar methods). This protocol is also open to other conditions whose basis is also thought to result from L-R problems. In all cases, the patients continue under the care of the referring physician. We anticipate a minor role of NIH researchers and genetic counseling services if subjects either do not have, or cannot afford, similar services in their local area.

This is not a treatment protocol. Our empiric ability to generate medically significant research results is limited by the extensive genetic and other etiologic heterogeneity. Therefore, this research is not a diagnostic study. At this stage of research, we are not sufficiently confident that our research results will have direct medical implications for research subjects.

Results that are of potential medical importance will be discussed with the primary physician who is (in most cases) a trained cardiologist (and/or medical geneticist). We will emphasize that these are only preliminary research findings, that they are not CLIA-approved, and must be disclosed to the patient or included in the medical record. Repeat testing in a CLIA-approved lab under another protocol would be required before the genetic information could be shared with the patient and family.

ELIGIBILITY:
* INCLUSION CRITERIA:

This research protocol is open to all participants with a known or suspected diagnosis of L-R axis malformations. Nationality or place of origin are not specific barriers to participation, provided that a blood or tissue sample can be safely sent by international FedEx (to be billed to our account).

Direct blood relatives (typicially parents, and occasionally affected siblings) of patients with L-R malformations are also eligible to participate.

EXCLUSION CRITERIA:

Anyone unwilling to provide informed consent (for themselves as adults, or on behalf of their children as minors) or assent.

Medical condition(s) are not in themselves reason for exclusion if in the judgment of the referring physician this would involve no more than minimal risk.

We generally review a brief clinical description from the referring physician about a potential research subject to determine that the subject is appropriate to enter into the study. We reserve the right to exclude cases that are clearly not related to our direct research interests (e.g. patients born with defects in the heart chambers, such as simple atrial or ventricular septal defects, would generally be excluded from this study).

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 900
Dates: Start 1999-12-13; Primary Completion 2006-11-27 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- National Human Genome Research Institute (NHGRI), 9000 Rockville Pike, Bethesda, Maryland, United States